CLINICAL TRIAL: NCT07317440
Title: Coenzyme Q10 as an Adjunct Therapy in Pediatric Community-Acquired Pneumonia
Brief Title: Coenzyme Q10 in Pediatric Community-Acquired Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Zaki Elmeazawy, Lecturer of pediatrics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1169/3/25
Record Dates: First submitted 2025-06-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 children with community acquired pneumonia will receive oral coenzymeQ10 (Experimental)
  Interventions: Drug: oral coenzymeQ10
- 60 children with community acquired pneumonia with the standard pneumonia treatment. (No Intervention)

INTERVENTIONS:
Drug: oral coenzymeQ10 — 60 children with community acquired pneumonia will receive oral coenzymeQ10 in capsule form at a dose of 100-200 mg/kg/day, as adjunct therapy to the usual pneumonia treatment till the recovery of the disease.
  Arms: 60 children with community acquired pneumonia will receive oral coenzymeQ10

SUMMARY:
The aim of this work is to assess the benefit of coenzyme Q10 supplementation, in addition to standard antibiotic and other supportive therapy, in the management of hospitalized children with community acquired pneumonia

ELIGIBILITY:
Inclusion Criteria:

* All children aged 2 months -18 years with community acquired pneumonia diagnosed by signs and symptoms of CAP including; chest pain, dyspnea, tachypnea, or abnormal auscultatory findings plus focal findings on chest x ray indicating community acquired pneumonia

Exclusion Criteria:

* Children with immunodeficiency, chronic lung disease, malignancy, congenital lung anomalies, underlying disorder impacting respiration i.e. genetic, metabolic, neuromuscular disorders, children with CHD affecting the pulmonary blood flow.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Normalization of respiratory rate | 3 days
Normalization of temperature | 3 days
Normalization of oxygen saturation | 3 days
Normalization of Feeding Behavior Assessed by Oral Intake Tolerance | 3 days
  Normalization of feeding refusal will be assessed by evaluating the child's ability to tolerate age-appropriate oral feeding without refusal over a 3-day observation period.
Serum C-Reactive Protein (CRP) Level | 5 days
  Blood samples will be collected, and CRP concentration will be expressed in milligrams per liter (mg/L).
Serum Lactate Dehydrogenase (LDH) Level | 5 days
  LDH concentration will be reported in units per liter (U/L) from venous blood samples.
Prognostic Nutritional Index | 5 days
Systemic Immune-Inflammation Index | 5 days
Serum C-Reactive Protein to Albumin Ratio (CRP/Albumin Ratio) | 5 days
  The serum C-reactive protein to albumin ratio (CRP/albumin ratio) will be calculated as a single composite outcome measure using laboratory values obtained from the same blood sample.
Time of clinical stability | 3-5 days

SECONDARY OUTCOMES:
Length of hospital stay | 10-21 days
Number of Participants Requiring Surgical Intervention | 21-30 days
  This outcome measures whether a participant undergoes any surgical intervention related to the study condition during the follow-up period. Surgical intervention is defined as any operative procedure performed under general or regional anesthesia, as documented in the medical record.
  The outcome will be recorded as a binary variable (Yes/No) for each participant and summarized as the number and proportion of participants requiring surgical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt